CLINICAL TRIAL: NCT05714787
Title: Opportunistic Screening for Vertebral Osteoporotic Fractures on Chest CT Scan Evaluation of Patients With Interstitial Lung Disease : COLIBRI Based Retrospective Study
Brief Title: Opportunistic Screening for Osteoporotic Vertebral Fractures in Patients With Diffuse Interstitial Lung Disease
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 23Rhumato01
Record Dates: First submitted 2023-01-20; First posted 2023-02-06 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Osteoporosis; Interstitial Lung Disease; Vertebral Fracture
MeSH Terms: conditions — Osteoporosis; Lung Diseases, Interstitial; Spinal Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Chest CT Scan examination — Double examination of chest CT scan on sagittal section after multiplanar reconstruction

SUMMARY:
It is well known that some chronic respiratory pathologies such as asthma or chronic obstructive pulmonary disease (COPD) are associated with an increased risk of osteoporosis, due to the pathology itself and the therapies implemented (per-os or inhaled corticosteroids). Osteoporosis leads to an increased risk of fragility fracture, with an increased morbidity and mortality associated with severe fractures such as vertebral fractures. Also, osteoporotic vertebral fractures often occur at the thoracolumbar hinge, resulting in worsening of the thoracic kyphosis. However, to the best of our knowledge, the prevalence of osteoporotic vertebral fractures measured by CT scan in patients with interstitial lung disease (ILD) is not known. For these patients who already have impaired respiratory function, the appearance of vertebral fractures could impact their management and worsen their prognosis (additional restrictive syndrome, difficulties in analgesics management because of respiratory contraindications, difficulties in wearing a corset, etc...). In this context, it appears interesting to define the prevalence of osteoporosis and osteoporotic vertebral fractures at the thoracic spine and the thoraco-lumbar hinge in a population of patients followed for ILD. So, the main objective of this study is to describe the prevalence of vertebral osteoporotic fractures in an overall cohort of patients with ILD.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years old ;
* Patients included in the COLIBRI database for ILD between January 2017 and January 2023 ;
* Patients with a chest CT scan performed at the Nice center university hospital.

Exclusion Criteria:

* Absence of a thoracic CT scan performed at Nice center university hospital
* Secondary vertebral fracture

Ages: 18 Years to 95 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients are from a cohort data base named COLIBRI which collected date about with intersititial lung disease, recruited in Pneumology Department in Centre hospitalier universitaire de Nice.
Sampling Method: Non-Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2017-01-23 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Presence or absence of vertebral fracture in the global cohort | 6 years
  a vertebral fracture is considered if a decrease in height of the vertebral plateau by more than 20 % on an examination of chest CT scan on sagittal section after multiplanar reconstruction is observed.

SECONDARY OUTCOMES:
Presence or absence of vertebral fracture in subgroups | 6 years
  a vertebral fracture is considered if a decrease in height of the vertebral plateau by more than 20 % on an examination of chest CT scan on sagittal section after multiplanar reconstruction is observed.
To compare bone mineral density in Hounsfield Unit of patients with or without at least one vertebral fracture. | 6 years
  Bone mineral density in hounsfield unit is evaluated by measuring trabecular attenuation in an ovoid region of interest on axial T12 section

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No
not scheduled